CLINICAL TRIAL: NCT01122615
Title: Phase I Trial of Sunitinib Plus Temsirolimus in Patients With Metastatic Renal Cell Cancer
Brief Title: Sunitinib Plus Temsirolimus in Patients With Renal Cell Cancer (RCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0037; NCI-2011-02066 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-07

CONDITIONS: Renal Cell Cancer; Kidney Cancer
Keywords: Kidney; metastatic renal cell carcinoma; RCC; Sunitinib; Sunitinib Malate; Sutent; Temsirolimus; Torisel
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib + Temsirolimus (Experimental): Sunitinib 12.5 to 50 mg orally (PO) daily x 14 days, 7 days off for 21 day cycle. Temsirolimus 6 to 25 mg intravenously (IV) over 30 minutes once weekly for 21 day cycle.
  Interventions: Drug: Sunitinib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Sunitinib — 12.5 to 50 mg orally (PO) daily x 14 days, 7 days off for 21 day cycle.
  Other Names: Sunitinib Malate; Sutent
Drug: Temsirolimus — 6 to 25 mg intravenously (IV) over 30 minutes once weekly for 21 day cycle.
  Other Names: CCI-779; Torisel

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of sunitinib and temsirolimus that can be given to patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
The Study Drugs:

Sunitinib is designed to block pathways that control important events (such as the growth of blood vessels) that are essential for the growth of cancer.

Temsirolimus is designed to block the growth of cancer cells, which may cause cancer cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the combination of sunitinib and temsirolimus based on when you joined this study. There will be 2 stages in this study.

Up to 5 dose levels of the study drug combination will be tested in Stage 1. Two (2) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

During Stage 2, different doses of the individual study drugs will be tested based on the highest tolerable combination dose that was found in Stage 1.

Study Drug Administration:

During each 3-week "study cycle," you will take sunitinib 1 time each day (either with or without food) for 2 weeks followed by 1 week of rest with no study drug.

You will receive temsirolimus by vein 1 time every week over 30-60 minutes. About 30 minutes before you receive temsirolimus, you will receive Benadryl (diphenhydramine) by vein over 30 minutes to help prevent side effects.

If you have any side effects from any of the drugs, tell the study doctor right away. The study doctor may then lower the dose or keep the dose level the same.

Study Visits:

Every week (right before you receive temsirolimus), blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of every cycle:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any drugs or treatments you may be receiving.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests (in addition to the weekly blood draw described above).

Every 6 weeks,:

* You will have the same imaging scans (CT and/or MRI scan) that you had at the screening visit. If you have stable disease after 2 scans, you will have these every 12 weeks.
* Blood (about 2 teaspoons) will be drawn to check your thyroid function.
* Urine will be collected for routine tests.

Blood Pressure Monitoring:

During the first 3 weeks of the study, your blood pressure will be checked weekly. This may be done at your local doctor's office. You should write down your blood pressure each time it is checked in a blood pressure journal that the study staff will give you and bring it with you when you see your doctor.

Length of Study:

You will remain on study for as long as you are benefiting. You will be taken off study if the disease gets worse or if you have intolerable side effects.

End-of-Study Visit:

After the last dose of study drug, you will have an end-of-study visit. At the end-of-study visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you may have experienced since your last visit.

This is an investigational study. Sunitinib and temsirolimus are both FDA approved and commercially available for the treatment of advanced kidney cancer. The use of the drugs in combination is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed metastatic RCC of any histological subtype
2. Patients must have evaluable disease
3. Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of these targeted agents in patients < 18 years of age, children will be excluded from this study. RCC in patients < 18 is exceedingly rare in any event.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 1
5. Patients must have adequate organ and marrow function within 14 days as defined below: a) Absolute neutrophil count >/= 1,500/µL; b) Platelet count >/= 100,000/µL; c) Hemoglobin >/= 9.0 g/dL (may be transfused to maintain or exceed this level); d) Total bilirubin </= 2.0 mg/dl; e) Albumin > 2.5 g/dL; f) Serum creatinine </= 2.0 mg/dl; g) AST (SGOT) and ALT (SGPT) </= 2.5 times the institutional upper limit of normal for subjects without evidence of liver metastases; h) AST (SGOT) and ALT (SGPT) </= 5 times the institutional upper limit of normal for subjects with documented liver metastases
6. Female patients of childbearing potential must have a normal serum beta human chorionic gonadotropin (beta-hCG) within 24 hours prior to beginning treatment on the study due to the possible teratogenic effect.
7. Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study
8. Patients must give written informed consent prior to initiation of study-related procedures. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
9. Patients must be able to swallow pills
10. Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

1. No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been definitively treated and disease free for 2 years. Patients with controlled brain metastases are eligible.
2. Patients must not be scheduled to receive another anticancer drug while on this study. Patients are permitted to be on concomitant bisphosphonates or megestrol acetate
3. Patients must not have had a stroke or TIA within 6 months
4. Patients must not have uncontrolled infections that could be worsened by anticancer therapy or interfere with this study
5. Patients must not have clinically significant cardiovascular disease, defined as myocardial infarction (or unstable angina) within 6 months, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia refractory to medical management, or peripheral vascular disease (Grade III or greater)
6. Patients must not have uncontrolled hypertension, defined as > 140/90 in either systolic or diastolic component (treatment of hypertension with medications is permitted)
7. Symptomatic peripheral vascular disease
8. Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breast-feeding should be discontinued if the mother is enrolled on this trial
9. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. In addition, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with some of these agents
10. Patients must not have a clinical history of coagulopathy or bleeding diathesis
11. Concomitant treatment with rifampin, St. John's wort, or the cytochrome p450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital) or CYP3A4 inhibitors is not recommended on this study.
12. Patients with significant baseline proteinuria defined as > grade 2 by screening U/A will be excluded if they have > 2 g protein by urine protein over creatinine (UPC) ratio
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
14. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device within 7 days prior to study enrollment
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
16. Non-healing wound, ulcer, or bone fracture
17. Known hypersensitivity to any component of sunitinib malate, or temsirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Sunitinib and Temsirolimus | 21 days
  Determination of MTD based on the occurrence of dose limiting toxicities (DLTs) during cycle one only after administration of study drugs on day one through day 21. All toxicity graded according to criteria of NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 3.0.

SECONDARY OUTCOMES:
Response Rate | 6 weeks
  Response and progression evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the index tumor lesions are used in the RECIST criteria. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LDof target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Nizar M. Tannir, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org